CLINICAL TRIAL: NCT07222839
Title: Exploring the Effect of Visually Immersive Video Education on Cardiothoracic Surgery Patients' Preoperative Anxiety and Postoperative Outcomes
Brief Title: Impact of Immersive Video Education on Cardiothoracic Surgery Anxiety and Outcomes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baptist Health South Florida (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2359886
Record Dates: First submitted 2025-09-23; First posted 2025-10-30 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-10

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention - Visually Immersive Video Education (Experimental): Participants receive visually immersive (virtual reality-designed) preoperative video education shown on a tablet that orients patients to the postoperative CVICU environment, equipment, and expected recovery processes. After viewing the video, the open-heart trained CVICU nurse provides opportunity for discussion, clarification, and questions. Assignment to this arm occurs during intervention weeks (Weeks 1-2 of each month, per protocol).
  Interventions: Behavioral: Visually Immersive Video
- Control - Standard Preoperative Education (Active Comparator): Participants receive standard preoperative education consisting of a basic verbal explanation of what to expect postoperatively on arrival to the CVICU, followed by opportunity for questions. Assignment to this arm occurs during control weeks (Weeks 3-4 of each month, per protocol).
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Behavioral: Visually Immersive Video — The patients watch a 5-minute visually immersive education video on what to expect postoperatively on arrival to the cardiovascular intensive care unit (CVICU) followed by the opportunity for discussion/explanation and questions.
  Arms: Intervention - Visually Immersive Video Education
Behavioral: Standard of Care — The patient receives a basic verbal explanation of what to expect postoperatively on arrival to CVICU followed by the opportunity for questions.
  Arms: Control - Standard Preoperative Education

SUMMARY:
The purpose of this quasi-experimental study is to examine the effect of visually immersive preoperative education on levels of anxiety and patient outcomes in patients undergoing cardiothoracic (open heart) surgery

ELIGIBILITY:
Inclusion Criteria:

* Inpatients and outpatients scheduled for elective cardiothoracic (open heart) surgery

Exclusion Criteria:

* Patients undergoing emergent cardiothoracic (open heart) surgery
* Patients with altered mental status
* History of mental health disorders (schizophrenia and bipolar disorder)
* Legally blind/complete blindness and hearing impaired (without hearing aids)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2027-01-15 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
Anxiety relief (self-report measure 1 - State-Trait Anxiety Inventory) | 30 minutes
  Patient's anxiety will be measured using the 20-item State-Trait Anxiety Inventory (STAI) (state scale only) (higher scores indicate higher anxiety), taken before and after preoperative education is received.
Anxiety relief (self-report measure 2 - Visual Analog Scale for Anxiety) | 30 minutes
  Patient's anxiety will be measured using the Visual Analog Scale for Anxiety (VAS-A), a slider scale of 0 - 100 is used to self-report anxiety (0 = not anxious and 100 = extremely anxious), taken before and after preoperative education is received.

SECONDARY OUTCOMES:
Anxiety relief (physiological measure 1 - blood pressure) | 30 minutes
  Blood pressure is measured before and after receipt of preoperative education. Increased anxiety may cause elevation of this physiological indicator.
Anxiety relief (physiological measure 2 - heart rate) | 30 minutes
  Heart rate is measured before and after receipt of preoperative education. Increased anxiety may cause elevation of this physiological indicator.
Anxiety relief (physiological measure 3 - respiratory rate) | 30 minutes
  Respiratory rate is measured before and after receipt of preoperative education. Increased anxiety may cause elevation of this physiological indicator.
Postoperative CVICU Outcome 1 - Length of Stay | Within 30 days after the patient is discharged from CVICU
  Patients' length of stay (# days) in the CVICU.
Postoperative CVICU Outcome 2 - Intubation Time | Within 30 days after the patient is discharged from CVICU
  Intubation time = Length of time the patient is on mechanical ventilation.
Postoperative CVICU Outcome 3 - Re-intubation | Within 30 days after the patient is discharged from CVICU
  Re-intubation after initial removal from mechanical ventilation (yes or no).
Postoperative CVICU Outcome 4 - Blood Sugar Regulation | Within 30 days after the patient is discharged from CVICU
  Blood sugar regulation = comparison of point-of-care blood sugar levels taken on postoperative day 1 and on the day of discharge from CVICU.

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Bermudez, PhD, RN, EBP-C, Study Chair — Baptist Health | Nursing & Health Sciences Research
Locations (1):
- South Miami Hospital, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No